CLINICAL TRIAL: NCT03539653
Title: The Effect of Gastric Antrum Ultrasonography on Early Stage of Enteral Nutrition in Critically Ill Patients.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kang Yan (Other)
Collaborators: Beijing Tsinghua Chang Gung Hospital (Other); Zhongda Hospital (Other); First Hospital of China Medical University (Other); Beijing Tongren Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor-Investigator, Kang Yan, Director, West China Hospital
Organization: West China Hospital (Other)
Other Study IDs: GUS
Record Dates: First submitted 2018-04-23; First posted 2018-05-29 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Critically Ill
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to investigate the effect of Gastric Antrum Ultrasonography on Early Stage of Enteral Nutrition in Critically Ill Patients.

ELIGIBILITY:
Inclusion Criteria:

All patients who need enteral nutrition (through the nose) in ICU ; the length of stay in ICU > 3 days;

Exclusion Criteria:

<18 years old; >90 years old; gastrointestinal surgery history； small blow nutrition； BMI>30kg/m2; pregnancy; prone position>4hours a day

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients in ICU who need enteral nutrition,and the length of stay in icu>3days
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
incidence of tube feeding intolerance during ICU | during ICU,an average of 7 days
  incidence of tube feeding intolerance during ICU，such as vomit，diarrhea，Bloating.

SECONDARY OUTCOMES:
gastric residual volume | during ICU,an average of 7 days
  gastric residual volume during ICU
nutrition indicators | through study completion,an average of 7 days
  nutrition indicators during ICU,such as prealbumin
the first clinical parameters of prognosis | through study completion,an average of 7 days
  incidence of regurgitation during enteral nutrition
the second clinical parameters of prognosis | through study completion,an average of 7 days
  ventilator-associated pneumonia
the third clinical parameters of prognosis | through study completion,an average of 7 days
  length of mechanic ventilation during ICU
the forth clinical parameters of prognosis | through study completion,an average of 7 days
  length of stay in ICU
the fifth clinical parameters of prognosis | through study completion,an average of 15 days
  hospital mortality
the sixth clinical parameters of prognosis | through study completion,an average of 7 days
  hospitalization costs during ICU

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Xu, M.D., Study Chair — Beijing Tsinghua Changgeng Hospital; Wei He, Study Chair — Beijing Tongren Hospital; Yi Yang, Study Chair — Zhongda Hospital; Bin Ouyang, Study Chair — The first affiliation hospital,Sun Yat-sen university; Ran Zhu, Study Chair — First Hospital of China Medical University
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

REFERENCES:
- [Background] McClave SA, Taylor BE, Martindale RG, Warren MM, Johnson DR, Braunschweig C, McCarthy MS, Davanos E, Rice TW, Cresci GA, Gervasio JM, Sacks GS, Roberts PR, Compher C; Society of Critical Care Medicine; American Society for Parenteral and Enteral Nutrition. Guidelines for the Provision and Assessment of Nutrition Support Therapy in the Adult Critically Ill Patient: Society of Critical Care Medicine (SCCM) and American Society for Parenteral and Enteral Nutrition (A.S.P.E.N.). JPEN J Parenter Enteral Nutr. 2016 Feb;40(2):159-211. doi: 10.1177/0148607115621863. No abstract available. PMID 26773077
- [Background] Warren M, McCarthy MS, Roberts PR. Practical Application of the Revised Guidelines for the Provision and Assessment of Nutrition Support Therapy in the Adult Critically Ill Patient: A Case Study Approach. Nutr Clin Pract. 2016 Jun;31(3):334-41. doi: 10.1177/0884533616640451. Epub 2016 Apr 12. PMID 27072854
- [Background] Sharma V, Gudivada D, Gueret R, Bailitz J. Ultrasound-Assessed Gastric Antral Area Correlates With Aspirated Tube Feed Volume in Enterally Fed Critically Ill Patients. Nutr Clin Pract. 2017 Apr;32(2):206-211. doi: 10.1177/0884533616681530. Epub 2016 Dec 16. PMID 28362573
- [Background] Liu Y, Gao YK, Yao L, Li L. Modified B-ultrasound method for measurement of antral section only to assess gastric function and guide enteral nutrition in critically ill patients. World J Gastroenterol. 2017 Jul 28;23(28):5229-5236. doi: 10.3748/wjg.v23.i28.5229. PMID 28811717
- [Background] Bisinotto FM, Pansani PL, Silveira LA, Naves AA, Peixoto AC, Lima HM, Martins LB. Qualitative and quantitative ultrasound assessment of gastric content. Rev Assoc Med Bras (1992). 2017 Feb;63(2):134-141. doi: 10.1590/1806-9282.63.02.134. PMID 28355374
- [Background] Van de Putte P, Perlas A. Ultrasound assessment of gastric content and volume. Br J Anaesth. 2014 Jul;113(1):12-22. doi: 10.1093/bja/aeu151. Epub 2014 Jun 3. PMID 24893784